CLINICAL TRIAL: NCT05135182
Title: Helicobacter Pylori Rescue Treatment Containing Tetracycline in Patients Allergic to Penicillin:a Prospective Randomized Controlled Study
Brief Title: Helicobacter Pylori Rescue Treatment in Patients Allergic to Penicillin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-SDU-QILU-G226
Record Dates: First submitted 2021-11-23; First posted 2021-11-26 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Eradication; Allergic; Penicillin; Tetracycline
MeSH Terms: interventions — Furazolidone; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- furazolidone-tetracycline-containing quadruple (Experimental): patients in furazolidone-tetracycline-containing quadruple group will receive vonoprazan fumarate 20mg po bid, tetracycline 500mg po qid , bismuth potassium citrate(Lizhudele) 220mg po bid, and furazolidone 100mg po bid for 14d
  Interventions: Drug: Furazolidone
- metronidazole-tetracycline-containing quadruple group (Active Comparator): patients in metronidazole-tetracycline-containing quadruple group will receive vonoprazan fumarate 20mg po bid,tetracycline 500mg po qid , bismuth potassium citrate(Lizhudele) 220mg po bid, and metronidazole 400mg po qid for 14d.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Furazolidone — Furazolidone-tetracycline-containing quadruple regimens
  Arms: furazolidone-tetracycline-containing quadruple
Drug: Metronidazole — metronidazole-tetracycline-containing quadruple regimens
  Arms: metronidazole-tetracycline-containing quadruple group

SUMMARY:
The purpose of this study is to assess and compare the effectiveness of furazolidone-tetracycline-containing and metronidazole-tetracycline-containing quadruple regimens for the rescue treatment of Helicobacter pylori infection inpatients allergic to penicillin.

DETAILED DESCRIPTION:
Helicobacter pylori(H.pylori), which infects about 50% of the global population,has been recognized as a main risk factor of multiple gastric pathologies,especially non-cardiac gastric cancer. Strongly evidence supports that H.pylori eradication is an effective approach to reduce the incidence of those pathologies.However,Helicobacter pylori eradication is a challenge in patients allergic to penicillin. Therefore, the investigators aim to assess and compare the effectiveness of furazolidone-tetracycline-containing and metronidazole-tetracycline-containing quadruple regimens for the rescue treatment of Helicobacter pylori infection in patients allergic to penicillin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with H. pylori infection.
* Patients with previous Helicobacter pylori eradication.
* Patients Allergic to Penicillin.

Exclusion Criteria:

* Patients treated with H2-receptor antagonist, PPI, bismuth and antibiotics in the previous 4 weeks.
* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer.
* Patients with known or suspected allergy to study medications.
* Currently pregnant or lactating.
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rates in 2 groups | 12 months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hosipital, Jinan, Shandong, China